CLINICAL TRIAL: NCT02873845
Title: Role of the Spouse/Partner of Persons Treated With Chemotherapy for Colon Cancer - Preliminary Validation of the Caregiver Objective Burden-Quality of Life (COBQoL) Questionnaire
Brief Title: Role of the Spouse/Partner of Persons Treated With Chemotherapy for Colon Cancer
Acronym: APPACH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LEJEUNE LaLigue 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- PATIENT: Patients with colon cancer
  Interventions: Other: Preliminary validation of the COBQoL questionnaire
- THE SPOUSE/PARTNER: The spouse/partner of patients with colon cancer
  Interventions: Other: Preliminary validation of the COBQoL questionnaire

INTERVENTIONS:
Other: Preliminary validation of the COBQoL questionnaire

SUMMARY:
Altered quality of life in patients with stage III or IV colon cancer is well known. At their sides, their spouse/partner must also cope with the suffering caused by the disease and the upheavals that it engenders, with the treatments, in the organization of their everyday life. The physical, emotional, social and financial impact of cancer in general and its treatment on care-givers has already been studied. However, there are no data concerning the "objective burden", that is to say the nature and the magnitude of the care weighing on the spouse of persons with colon cancer. Objective is to develop and validate a questionnaire that can be completed by the spouse/partner of patients with stage III or IV colon cancer so as to evaluate the burden of the disease in everyday life. It will allow medico-social professionals to identify spouses/partners in difficulty and the needs of patients so as to offer the best support.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients:

Men or women :

* able to understand written and spoken French ;
* Who have been informed about the study;
* with stage III or IV cancer of the colon or recto-sigmoid junction (Code C18 and C19 of the ICD 10), operated or not with curative intent; treated with chemotherapy in one of the study centres (adjuvant or 1st-line chemotherapy or palliative chemotherapy);
* Currently living with a spouse or partner;
* Who has consented to his/her spouse/partner taking part in the study.

Inclusion criteria for the spouse/partner:

Men or women:

* able to understand written and spoken French ;
* Who have been informed about the study; living at the home of the spouse/partner;
* Able to take part in an interview of approximately one hour;
* Who has provided consent to take part in the study.

Exclusion Criteria:

Exclusion criteria for patients:

Men or women :

* Under guardianship;
* With a severe disease resulting in a major handicap;
* With severe mental retardation affecting ability to understand;
* With rectal cancer;
* with stage I or II cancer of the colon or recto-sigmoid junction;
* with a history of treated cancer (colorectal or other);
* with another cancer under treatment

Exclusion criteria for the spouse:

Men or women:

* Under guardianship;
* With a severe disease resulting in a major handicap;
* With severe mental retardation affecting ability to understand

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their spouse/partner
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective burden score in the dimensions of the COBQoL questionnaire with good psychometric properties | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France